CLINICAL TRIAL: NCT03671252
Title: Prospectively Randomized Control Clinical Trial of FOLFOXIRI Preoperative Chemotherapy Alone on Rectal Cancer in Local Advance Comparing to Oral Capecitabine Combined With Long-term Radiation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, president of SunYat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAVORE Trial
Record Dates: First submitted 2018-08-28; First posted 2018-09-14 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol; XELOX; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group 1 (Experimental): Patient will receive FOLFOXIRI regimen every two weeks for 4-6 cycles within 2-3 months.Two weeks after completing 3 and 6 cycles of FOLFOXIRI regimen,patients will have two efficacy evaluations according to RECIST criteria and toxicity evaluation .If the tumor is defined as no progression without severe toxicity at the first efficacy evaluation, the rest of 3 cycles of FOLFOXIRI regimen will be performed.If it is defined as progression of primary tumor or it is defined as progression of primary tumor and MRF(+)at the second efficacy evaluation,patients are assigned into active comparator group. If distant metastasis occurred during chemotherapy, patients are treated according to the guidelines for metastatic colorectal cancer.Chemotherapy is initiated at 3-4 weeks after R0 resection. XELOX regimen is performed post-operatively (about 4-6 cycles). If postoperative pathology confirmed as positive margin, postoperative chemoradiotherapy was given.
  Interventions: Drug: FOLFOXIRI; Drug: XELOX; Other: Chemoradiotherapy; Procedure: TME operation; Procedure: efficacy evaluation
- Active Comparator:Group 2 (Active Comparator): The patients are scheduled to receive chemoradiotherapy. After 5 weeks from the end of chemoradiotherapy, patients will have a efficacy evaluation according to RECIST criteria. If the tumor is defined as CR、PR or SD, and the TME operation is conducted within 5-10 weeks after chemoradiotherapy completion. If tumor is defined as progressive disease with the possibility of R0 resection, the operation was also conducted within 5-10 weeks after chemoradiotherapy . If tumor is defined as progressive disease without possibility of R0 resection, the palliative chemotherapy was performed . If distant metastasis occurred during chemoradiotherapy, patients are treated according to the guidelines for metastatic colorectal cancer. Adjuvant chemotherapy of XELOX is performed post-operatively (about 4-6 cycles).
  Interventions: Drug: XELOX; Other: Chemoradiotherapy; Procedure: TME operation; Procedure: efficacy evaluation

INTERVENTIONS:
Drug: FOLFOXIRI — Irinotecan165 mg/m2、Oxaliplatin85 mg/m2、Left-calcium leucovorin 200mg/㎡，Intravenous infusion，first day. Then, 5-FU 1600 mg/m2/d×2 continuous intravenous infusion（total 3200 mg/m2，infusion 46 hours）in the next two days. Repeat every 14 days.
  Arms: Experimental: Group 1
Drug: XELOX — XELOX consisting of 130 mg/m2 oxaliplatin administered intravenously on day 1 and 1,000 mg/m2 capecitabine administered orally twice daily on days 1-14 for a 3-week cycle.
Other: Chemoradiotherapy — Chemotherapy: oral capecitabine（1650 mg/m2）twice daily during radiotherapy without weekend breaks.
  Radiation: Radiation therapy is administered via intensity-modulated radiation therapy (IMRT) with a linear accelerator, 6MV-X ray. The patients are scheduled to receive a GTV expanding 6mm to form PTV1 and CTV expanding 6mm to form PTV2. The dose of PTV1 is 50Gy/25 times for 35 days and the dose of PTV2 is 45Gy/25 times for 35 days. Patients were treated in consecutive days per week for a total of 5 weeks.
Procedure: TME operation — TME operation
Procedure: efficacy evaluation — chest/ abdominal CT、pelvic nuclear magnetic resonanceimaging、transrectal ultrasonography

SUMMARY:
Preoperative radiation and chemotherapy is the standard treatment for local advanced rectal cancer. The addition of oxaliplatin to capecitabine combined with radiotherapy does not improve local control and long-term survival. Most importantly,chemoradiotherapy significantly increased surgical complication and poor long-term quality of life .In the absence of effective measures of predicting chemo-sensitivity, there is considerable risk of using any two-drug regimen for neoadjuvant therapy. Simultaneous use of the three chemotherapeutic drugs may be able to reduce the likelihood of resistance to both dual drug regimen and single drug regimen. The purpose of this study is to compare the efficacy and safety of three chemotherapeutic regimen known as FOLFOXIRI (the drug 5-fluorouracil, oxaliplatin, Irinotecan) with standard radiotherapy combined with capecitabine in neoadjuvant therapy for local advanced rectal cancer. The drugs in the FOLFOXIRI regimen are all FDA(Food and Drug Administration) approved and have been used routinely to treat patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Outline: This is a multicenter,prospectively,randomized control ,phase III clinical study.Patients are stratified according to the distance from the tumor to the anal margin（≤5cm，>5cm） and randomized to 1 of 2 treatment regimen.Patients will receive full supportive care while on this study.

Objectives：

Primary: To compare neoadjuvant chemotherpay of FOLFOXIRI with conventional capecitabine single-agent radiotherapy in local advanced rectal cancer with respect to 3-year disease free survival rate (DFS) .

Secondary:

1. To compare postoperative 3-year local recurrence rate, 3-year distance metastasis free survival rate, 3-year overall survival between neoadjuvant FOLFOXIRI with capecitabine single-agent radiotherapy groups.
2. To compare R0 Resection rate and surgical complication between the two groups.
3. To evaluate the tumor regression grade(TRG) between the two groups.
4. To evaluate the adverse event profile and Long term quality of life between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1）Age: 18 to 75 years old;
* 2）Histological diagnosis of rectal adenocarcinoma;
* 3）Distance form anal margin ≤ 5cm: cT3-4aN + M0, there is no distant metastasis, lymph node positive, or the tumor breaking through the muscular layer, no invasion of the adjacent organs , positive MRF, it is estimated that R0 resection can be performed;
* 4）From the anal margin>5cm: cT3c-4aN+M0, there is no distant metastasis, lymph node positive, or the tumor breaking through the muscular layer with invading the mesorectum more than 5mm, no invasion of the adjacent organs, positive MRF, it is estimated that R0 resection can be performed;
* 5）Preoperative staging method: All patients undergoing anal examination, high-resolution MRI and/or EUS for preoperative staging. The diameter of parenteral lymph node ≥10mm, lymph node shape or the MRI characteristics is consistent with typical lymph node metastasis. If combined with EUS, the material should be submitted to the central assessment team for judgment when there is a contradiction in the staging method. Preoperative chest and abdomen CT, pelvic MRI are used for excluding distant metastasis;
* 6）Confirmed as the lower edge of tumor is located within 12 cm from the anal margin by MRI examination
* 7）There is no signs of intestinal obstruction, or obstruction of intestinal after treating with proximal colostomy has been relieved;
* 8）Patients did not previously receive rectal surgery, chemotherapy or radiation therapy , biological treatment , except for endocrine therapy;
* 9）ECOG Performance Status :0-1
* 10）Life expectancy: more than 2 years;
* 11）Laboratory values：Hematology: white blood cell count>4000/mm3; Platelet count>100000/mm3; Hemoglobin >10g/dL; Liver function: SGOT and SGPT < 1.5 upper limit of normal(ULN); Bilirubin< 1.5mg/dL; Renal function :Creatinine <1.8mg/dL.

Exclusion Criteria:

* 1）Tumor invasion of surrounding tissue organs (T4b) by preoperative staging assessment;
* 2）Obturator lymph node metastasis;
* 3）Arrhythmia requires treatment with antiarrhythmia (except for beta-blockers or digoxin), symptomatic coronary artery disease, myocardial ischemia (myocardial infarction within the last 6 months) or congestive heart failure exceeding NYHA class II;
* 4）Severe hypertension with poor control;
* 5）History of HIV infection or active phase of chronic hepatitis B or C infection with high copy viral DNA;
* 6）Other active serious infections according to NCI-CTC version 4.0;
* 7）There is preoperative evidence for distant metastasis outside pelvis;
* 8）Cachexia and organ function decompensation
* 9）History of pelvic or abdominal radiotherapy;
* 10）Multiple primary cancer;
* 11）Patients with epilepcy requiring treatment ( steroids or antiepileptic treatment);
* 12）History of other malignant tumors within 5 years, except for cured cervical carcinoma in situ or skin basal cell carcinoma;
* 13）Drug abuse and medical, psychological or social conditions interfering patient participation in research or the evaluation of research results;
* 14）Any allergy to clinical research drugs or any drugs associated with this study;
* 15）Any unstable condition or condition that may endanger safety and compliance of patients;
* 16）Pregnancy or the lactating female without adequate contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Estimated)
Dates: Start 2018-11-16 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | up to 5 years
  3-year disease free survival was defined as the interval from randomization to disease local recurrence and distance metastasis, death, or the last follow-up within 3 years. Patients without any event (metastasis or death) at the last follow-up date were regarded as random censoring.

SECONDARY OUTCOMES:
3-year local recurrence rate | up to 5 years
  3-year disease local recurrence was defined as the interval from randomization to local recurrence, death, or the last follow-up within 3 years. Patients without any event (local recurrence or death) at the last follow-up date were regarded as random censoring.
3-year distance metastasis free survival rate | up to 5 years
  3-year distance metastasis was defined as the interval from randomization to distance metastasis, death, or the last follow-up within 3 years. Patients without any event (distance metastasis or death) at the last follow-up date were regarded as random censoring.
5-year overall survival rate | up to 5 years
  5-year overall survival was defined as the interval from the date of randomization until death of any cause or the last follow-up within 5 years.
R0 Resection rate | up to 5 years
  Percentage of included patients who were performed radical tumor resection among total included patients
Surgical complication | up to 5 years
  Surgical complication including anastomotic leakage , anastomotic stricture , intestinal obstruction , postoperative pelvic bleeding, and poor wound healing.
Tumor regression grade (TRG) | up to 5 years
  The tumor regression grade(TRG) were assessed using the Mandard TRG system.
Number of Adverse events | up to 5 years
  Treatment related adverse events were evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (CTCAE4.0)
Long term quality of life | up to 5 years
  Long term quality of life were assessed by European organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ C30)

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Cancer center of Sun Yat-sen University, Guangzhou, Guangdong
  - Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong